CLINICAL TRIAL: NCT01135277
Title: Immune Suppression and Ventilator Associated Pneumonias
Acronym: iVAP
Status: Completed | Type: Observational
Sponsor: Matthew Exline (Other)
Responsible Party: Sponsor-Investigator, Matthew Exline, Assistant Professor Clinical, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2009H0165
Record Dates: First submitted 2010-05-26; First posted 2010-06-02 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood Bronchoalveolar lavage fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Sepsis: Patients who have been diagnosed with Sepsis within 24 hours of admission
- Non-Septic: Patients who have not been diagnosed with sepsis within 24 hours of admission

SUMMARY:
Patients in the ICU are already predisposed to nosocomial infections, which are both costly and potentially life threatening, and it appears that the immune paralysis of sepsis may put these patients at greater risk for secondary infections, though this has not been proven conclusively. One measure of this sepsis-induced immune suppression is monocyte deactivation. The investigators hypothesize that, as a cornerstone of the monocytic innate immune response to infection, the inflammasome is critical to monocyte function during sepsis.

DETAILED DESCRIPTION:
Sepsis is a systemic inflammatory response to a severe infection. Despite the high incidence and societal costs of sepsis, the mechanism by which it kills remains unclear. The pathophysiology of sepsis is not completely understood, but many investigators now believe that sepsis induces a prolonged state of immune suppression. This study will attempt to quantify the degree of immune suppression during the first 5 days of sepsis by measuring the immune function of peripheral blood monocytes and the inflammasome constituent proteins in peripheral blood monocytes and alveolar macrophages.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years.
2. Have consensus criteria for sepsis (infection plus two of four systemic inflammatory response syndrome [SIRS] signs [tachycardia, tachypnea, fever or hypothermia, leukocytosis or leukopenia]) and a known or suspected infection for SEPTIC arm.

   * Patients without criteria for sepsis will be eligible for CONTROL arm. Patient must consent to have blood drawn within 24 hours of initiation of mechanical ventilation (for CONTROL arm) and 24 hours of new episode of sepsis to be eligible (for SEPTIC arm).

Exclusion Criteria:

1. Consent not available or declined
2. Prisoner
3. Died before blood collected
4. Onset of sepsis more than 24 hours prior to transfer to OSUMC,mechanical ventilation greater than 24 hours
5. Anticipation of less than 24 hours of mechanical ventilation by primary team
6. Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be open to males and females, 18 years or older, who spend at least one day on mechanic ventilation in the Ohio State University Medical Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2010-02; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Immune suppression during the recovery from critical illness is greater in severe sepsis patients compared to non-septic patients. | Day 1
  Blood and BAL fluid will be collected at Day 1
Immune suppression during the recovery from critical illness is greater in severe sepsis patients compared to non-septic patients. | Day 3
  Blood and BAL fluid will be collected at Day 3
Immune suppression during the recovery from critical illness is greater in severe sepsis patients compared to non-septic patients. | Day 5
  Blood and BAL fluid will be collected at Day 5

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Exline, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States